CLINICAL TRIAL: NCT00000747
Title: An Open-Label, Pilot Study to Evaluate the Development of Resistance to Nevirapine (BI-RG-587) in HIV-Infected Patients With CD4 Cell Count >= 500/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Boehringer Ingelheim (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 208; BI 00947
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Drug Resistance; AIDS-Related Complex; Antiviral Agents; Nevirapine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
Primary: To evaluate the rate of development of resistance to nevirapine in HIV-1 infected individuals. To evaluate safety of nevirapine in HIV-1 infected individuals with CD4 counts greater than or equal to 500 cells/mm3.

Secondary: To evaluate the effect of nevirapine on surrogate markers. The anti-HIV agent nevirapine is associated with rapid emergence of resistance when administered alone or in combination with zidovudine to HIV-infected patients with CD4 counts <= 400 cells/mm3. In persons with less advanced HIV disease and less viral burden, the emergence of resistance may be delayed, thus permitting evaluation for beneficial effect in a population where there is currently no established therapy.

DETAILED DESCRIPTION:
The anti-HIV agent nevirapine is associated with rapid emergence of resistance when administered alone or in combination with zidovudine to HIV-infected patients with CD4 counts <= 400 cells/mm3. In persons with less advanced HIV disease and less viral burden, the emergence of resistance may be delayed, thus permitting evaluation for beneficial effect in a population where there is currently no established therapy.

Ten patients receive nevirapine daily for 12 weeks. After 12 weeks of therapy, patients in whom resistance was not evident at week 4 and who have an adequate safety profile continue receiving nevirapine for an additional 12 weeks. Clinical and immunological assessments are performed at weeks 4, 8, 12, 16, 20, and 24. Virological assessments are performed at week 24 only. If 50 percent of patients develop resistance at any time, the study is discontinued.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Positive serum antibody to HIV-1 by ELISA or Western blot.
* CD4 count >= 500 cells/mm3 within 2 months prior to study entry, with two additional counts averaging >= 450 cells/mm3 at baseline and on study day 0 (taken at least 48 hours apart).
* No AIDS-defining disease.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* More than four loose stools per day.
* Participation in other experimental trials including vaccine trials.

Concurrent Medication:

Excluded:

* Other approved or investigational antiretroviral agents, other investigational agents, or vaccines.
* Glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulants.
* Digitoxin.
* Valproic acid.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Phenobarbital and other barbiturates.

Excluded 4 hours before or after a nevirapine dose:

* Antacids (particularly those containing calcium carbonate).
* H-2 blockers, carafate, cholestyramine resin, alcohol and alcohol-containing substances, and benzodiazepines (e.g., diazepam, triazolam).

Patients with the following prior conditions are excluded:

* History of clinically important disease other than HIV infection.

Prior Medication:

Excluded within 1 month prior to study entry:

* Any immunosuppressive, immunomodulatory, or cytotoxic treatment.

Use of drugs or alcohol sufficient to impair compliance with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Primary Completion 1994-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richman D, Study Chair
Locations (1):
- UCSD, San Diego, California, United States

REFERENCES:
- [Background] Havlir D. An open-label pilot study to evaluate the development of resistance to nevirapine (BI-RG-587) in HIV-infected patients with CD4 cell count > or = 500/mm. ACTG 208 Study Team. Int Conf AIDS. 1993 Jun 6-11;9(1):470 (abstract no PO-B26-2009)
- [Background] Havlir D, McLaughlin MM, Richman DD. A pilot study to evaluate the development of resistance to nevirapine in asymptomatic human immunodeficiency virus-infected patients with CD4 cell counts of > 500/mm3: AIDS Clinical Trials Group Protocol 208. J Infect Dis. 1995 Nov;172(5):1379-83. doi: 10.1093/infdis/172.5.1379. PMID 7594683